CLINICAL TRIAL: NCT06555926
Title: Effect of Acupressure on Carpal Tunnel Syndrome in Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant Hesham Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005286
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Acupressure; Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): The pregnant women will receive acupressure and advice for 12 weeks
  Interventions: Other: Acupressure; Other: advices for relieving carpal tunnel syndrome
- Advice group (Active Comparator): The pregnant women will receive advice only for 12 weeks
  Interventions: Other: advices for relieving carpal tunnel syndrome

INTERVENTIONS:
Other: Acupressure — The pregnant women will receive acupressure on the (Pc-6/Lung-7 )acupoints one minute for each point with 3 repetitions on both side( about 30minutes /session),2 times per week in addition to advices for 12 weeks.
  Arms: Acupressure group
Other: advices for relieving carpal tunnel syndrome — The pregnant women will receive advices for 12 weeks as follows:
  * Avoid heavy lifting.
  * Avoid repetitive tasks.
  * Sit on chairs with armrests and elevate affected hand on the armrest
  * Avoid sleeping on the side of the affected hand.
  * Keep the wrist in a neutral (straight) position.
  * Avoid positions of full flexion and extension.
  * Reduce general swelling by:
    * eating less salty food .
    * elevating legs when sitting .
    * wearing compression garments.
  * Apply cold water over the wrist.

SUMMARY:
This study will be conducted to investigate the effect of acupressure on carpal tunnel syndrome in pregnant women.

DETAILED DESCRIPTION:
The pregnant women are more prone to develop carpal tunnel syndrome because they retain more fluid during the later stages of their pregnancies. The more fluid retained , the more swelling occurs , squeezing the nerves that run through the hand and finger. Also most women who experience pain, numbness and tingling in the hand for the first time due to pregnancy have no idea that they have carpal tunnel syndrome.

Given the importance of treating CTS and preventing the limitations caused by this syndrome, and since it can turn into a debilitating disease if left untreated, acupressure can be recommended as a safe and noninvasive technique for reducing the severity of clinical symptoms.

Till now, there is no previous studies explored the effect of acupressure on carpal tunnel syndrome in pregnant women. So, this study will be conducted to provide new information about the efficacy of acupressure in management of carpal tunnel syndrome in pregnant women, which will help such pregnant women to overcome this problem and will add new evidence to the field of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are clinically diagnosed as having carpal tunnel syndrome .
* Their age will be ranged from 20 to 35years old.
* Their body mass index will not exceed 30kg/m2.
* All of them are in their 3rd trimester of pregnancy.(28-40weeks)
* All of them suffer from mild and moderate CTS.
* Degree of carpal tunnel pain will be 2 or more on Visual Analogue scale.

Exclusion Criteria:

* Dermatological abnormalities in the skin of acupionts.
* Internal fixation at the area of acupressure application.
* Smokers .
* Metabolic diseases such as Diabetes mellitus.
* Females who had history of fracture or trauma to the hand .

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain severity | 12 weeks
  The pain intensity will be assessed for all participants in both groups before and after treatment through VAS. It is a 10 cm horizontal line on which the participant's pain intensity will be represented by a point between the extremes of "no pain at all" and "worst imaginable pain". Each participant will be asked to mark a point on a VAS line between the extremes that related to her current pain intensity
median nerve conduction study | 12 weeks
  Computerized Electromyography (Dantce): ATOENINIES neuro screen system will be used to perform median nerve conduction study before and after the treatment program for all participants in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Azza Nashed, professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol